CLINICAL TRIAL: NCT06011226
Title: Development of a Patient-reported Outcome Measure for Chiari Malformation and Syringomyelia
Acronym: BCS-score
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP220733; 2022-A01816-37 (Other: IDRCB)
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-07

CONDITIONS: Syringomyelia; Chiari Malformation
Keywords: Syringomyelia; Chiari Malformation; patient-reported outcome measure
MeSH Terms: conditions — Syringomyelia; Arnold-Chiari Malformation | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1: development of the questionnaire: development of the patient reported outcome: The strategy consists of four phases:
  1. structured litterature review
  2. Group of experts: identification of the main areas to be covered by the questionnaire in order to draw up the focus group moderation guide
  3. focus groups: A discussion session will explore patient symptomatology, the functional impact of the disease, quality of life and the problems faced by patients from their point of view.
  Interventions: Other: focus groups
- Phase 2: pilot phase: Once the initial version of the self-questionnaire has been developed, it will be tested on a group of 40 patients with either Chiari malformation with syringomyelia (n = 20), isolated Chiari malformation (n = 10) or isolated syringomyelia (n = 10), managed by the CRMR C-MAVEM at Bicêtre Hospital.
  Interventions: Other: questionnaire
- Phase 3: national testing of the questionnaire: the 3rd phase will be submitted to the Human Subjects Protection Review Board according to the progression of the first two phases.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: focus groups — A dozen patients with Chiari malformation and syringomyelia (n = 4) or isolated Chiari malformation (n = 4) or isolated syringomyelia (n = 4) will be brought together in at least two focus groups. Each focus group will include 5 to 8 patients and will last approximately 1 to 2 hours. The focus groups will be recorded (audio only, no personal data will be collected during these sessions) and will be conducted in the presence of a neurosurgeon and a psychologist, who will moderate the session.
  Groups: Phase 1: development of the questionnaire
Other: questionnaire — developed questionnaire will be proposed to the patients in phase 2 and 3
  Groups: Phase 2: pilot phase; Phase 3: national testing of the questionnaire

SUMMARY:
Chiari malformation corresponds to the herniation of cerebellar tonsils into the foramen magnum resulting in obstruction of cerebrospinal fluid circulation, which may eventually lead to the formation of an intramedullary cavity called syringomyelia.

Chiari and syringomyelia can be responsible of variable symptoms, based on which neurosurgeons might propose surgical treatment. Yet, there is no properly developped and validated patient reported outcome measure (PROM) to assess the clinical severity of Chiari malformation and/or syringomyelia. The lack of such evaluation tool is a major issue to determine the optimal therapeutic strategy and to achieve a standardized and reproducible follow-up.

DETAILED DESCRIPTION:
Chiari malformation corresponds to the herniation of cerebellar tonsils into the foramen magnum resulting in obstruction of cerebrospinal fluid circulation, which may eventually lead to the formation of an intramedullary cavity called syringomyelia.

Chiari and syringomyelia can be responsible of variable symptoms, based on which neurosurgeons might propose surgical treatment. Yet, there is no properly developped and validated patient reported outcome measure (PROM) to assess the clinical severity of Chiari malformation and/or syringomyelia. The lack of such evaluation tool is a major issue to determine the optimal therapeutic strategy and to achieve a standardized and reproducible follow-up. The project will consist of two successive phases: a survey design of the questionnaire with small selected groups of patients; a monocentric pilot study on a limited population; The purpose of the development study is to produce a first version of the PROM based on proposed items written by experts and tested with volunteer patients (n = 10-20) within the framework of " focus groups" followed by cognitive debriefings. These items will explore various dimensions of the functional impact of Chiari malformation and syringomyelia (pain, motor disability, sphincter disorders, quality of life, etc.). The pilot study will test this 1st version of the questionnaire on a limited population of patients (n = 40) within the CRMR C-MAVEM of Bicêtre hospital to produce a final version. This work will be supplemented subsequently by a multicenter study allowing to validate a simple and reproducible evaluation tool in order to ensure the follow-up of patients with a Chiari malformation and/or syringomyelia and to measure surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to all subjects included in the study

* Age > 18 years
* Subject understanding French Patients included in Phase I
* Subject with signed informed consent Patients included in phase II
* Patient not opposed to study participation

Patients Chiari only group:

* Isolated descent of cerebellar tonsils > 5 mm below McRae's line (no associated syringomyelia)

Patients syringomyelia only group:

* Presence of an intramedullary fluid cavity secondary to circulatory disturbance of cerebrospinal fluid of non foraminal origin (no Chiari)

Patients Chiari with Syringomyelia group:

* Presence of Chiari malformation (tonsils > 5 mm below McRae's line) AND foraminal syringomyelia.

Exclusion Criteria:

* Insufficient command of French
* Minor or protected adult (guardianship, curatorship, safeguard of justice)
* Diagnosis of Chiari and/or syringomyelia not proven by an MRI scan
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The development of a questionnaire for self-assessment of the clinical impact of a pathology necessarily requires the involvement of the patients concerned. In particular, it is important that the clinical heterogeneity of the patients concerned is represented. The study population will therefore be patients with Chiari malformation, whether or not they have associated syringomyelia, and whether or not they have foraminal syringomyelia. They will be recruited via neurosurgical centers belonging to the C-MAVEM (Chiari, syringomyelia and vertebro-medullary malformations) network of rare disease reference centers for Chiari malformations and syringomyelia, and with the help of the main patient association (APAISER).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
development of metrologic and psychometric features of a patient-reported outcome measure (Bicêtre Chiari and Syringomyelia score - BCS score) | throughout the study (an average of 26 months)
  Development of metrologic and psychometric features of a patient-reported outcome measure (Bicêtre Chiari and Syringomyelia score - BCS score) for evaluating functional severity of Chiari malformation and/or syringomyelia
validation of metrologic and psychometric features of a patient-reported outcome | throughout the study (an average of 26 months)
  validation of metrologic and psychometric features of a patient-reported outcome measure (Bicêtre Chiari and Syringomyelia score - BCS score) for evaluating functional severity of Chiari malformation and/or syringomyelia

CONTACTS AND LOCATIONS:
Overall Officials: Steven KNAFO, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Hôpital Bicêtre
Locations (1):
- Hôpital Bicêtre - Service de Neurochirurgie - CRMR C-MAVEM, Le Kremlin-Bicêtre, France